CLINICAL TRIAL: NCT03998644
Title: A Study Focused on the Host and Microbiome of Colorectal Cancer Patients
Brief Title: Colorectal Cancer Associated Host and Microbiome Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, Professor, Shanghai 10th People's Hospital
Other Study IDs: CCAHMS
Record Dates: First submitted 2016-12-26; First posted 2019-06-26 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy: Subjects without colorectal disorders.
- precancerous: Subjects with risk factors that may contribute to the carcinogenesis.
- colorectal cancer: Patients who were identified by standard procedures to suffer with colorectal cancer.

INTERVENTIONS:
Other:

SUMMARY:
Recruit of healthy, precancer and colorectal cancer patients and record necessary information of demographic and also other messages. All the volunteers were asked to provide samples including stool, blood, urine and tissues. This protocol is performed with the permission of the ethics committee and all the participants were provided with informed consent.

DETAILED DESCRIPTION:
Healthy subjects, precancer patients identified by colonoscopy or colonoscopy history and colorectal cancer patients identified by two independent pathologists will be enrolled. The demographic message including age, weight, height, drug history, family history of all participants will be recorded. Blood, stool and urine samples will be collected of all subjects. Tumor and adjacent tissue samples of colorectal cancer and precancer patients were collected, as well as normal tissue of healthy subjects.

ELIGIBILITY:
Inclusion Criteria

1. individuals who were clear and signed the informed consent.
2. Male and female.
3. Age >18

Exclusion Criteria:

1. Any one who can not provide accurate information.
2. Any one who denies the study.
3. Younger than 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three different groups were created by healthy volunteers, precancerous and colorectal cancer patients. The information of these individuals will be analyzed and some conclusions will be drawn.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota structure and function difference between colorectal cancer, precancer and healthy controls | average of 5 years
  The results were based on the 16S rRNA metagenomic sequencing.

SECONDARY OUTCOMES:
Metabolic difference of blood samples between colorectal cancer, precancer and healthy controls | average of 5 years
  The metabolites of the blood samples by LC-MS will be detected.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No